CLINICAL TRIAL: NCT04411095
Title: The Effect of the Release of the Intrathoracic Fascia on Thoracic Rotation Mobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Academy of Osteopathy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: InternationalIAO
Record Dates: First submitted 2020-04-22; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Fascia; Inflammation; Thoracic; Rotation
MeSH Terms: conditions — Fasciitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stretching of intrathoracic fascia (Experimental): A technique will be used to stretch the intrathoracic fascia. The subject lies in his/her back, and a flexion of the upper cervical spine is combined with a retraction movement of the lower cervical and upper thoracic spine, this in combination with inspiration.
  Interventions: Other: Measuring thoracic rotation mobility
- Test without stretching (Placebo Comparator): A placebo technique is performed by positioning the hands of the therapist on the thorax without pressure or performing a technique. Similar as the stretching technique, a deep inspiration is performed by the patient, for each of the intrathoracic cilinders. This without performing a retraction of the lower cervical and upper thoracic spine.
  Interventions: Other: Measuring thoracic rotation mobility

INTERVENTIONS:
Other: Measuring thoracic rotation mobility — Measuring the thoracic rotation mobility with a goniometer, from a standardized position

SUMMARY:
Testing the effect of a specific stretch technique versus sham treatment, to objectify the influence of that specific technique on thoracic rotation mobility.

DETAILED DESCRIPTION:
Subjects in the experimental group will undergo a technique for stretching the intrathoracic fascia. Before and after, a measurement will be performed with a goniometer, to see if there is a difference in thoracic rotation mobility.

Subjects in the placebo group get a different technique, where the hands of the therapists are simply placed on the thorax, but no manoeuvre will be performed. Before and after, there is a measurement in thoracic rotation mobility.

Data will be compared and statistical analyse will be done to see of there is a difference in rotation. So the hypothesis that stretching intrathoracic fascia has an effect on thoracic rotation mobility, will be accepted or rejected.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the age of 18 and 65
* Both men and women

Exclusion Criteria:

* Structural disease of cervical or/and thoracic spine and/or head and/or thorax
* Acute mobility restriction of cervical and/or thoracic spine
* Acute and/or intense pain
* A history of trauma and/or operation on cervical and/or thoracic spine
* Treatment for cancer like chemo or radiation
* Baby's and children
* Elderly people

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Change in thoracic rotation mobility | Before and immediately after the test
  Change from baseline rotation, left and right, to rotation immediately after the test

CONTACTS AND LOCATIONS:
Overall Officials: IAO Administration, Study Director — The International Academy of Osteopathy
Locations (1):
- Practice for fysiotherapy and osteopathy, Scherpenheuvel, Vlaams-brabant, Belgium

IPD SHARING:
Plan to Share IPD: No